CLINICAL TRIAL: NCT06275802
Title: The Effect of Nutrition Education Interventions on Nutritional Status, Nutritional Habits and Eating Behaviors in Adolescents
Brief Title: The Effect of Nutrition Education Interventions for Adolescents
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Rana Nagihan AKDER, Research Assistant, Ege University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 22-5.1T/2
Record Dates: First submitted 2023-01-18; First posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Nutrition, Healthy; Nutrition Disorders in Adolescence; Eating Habit; Eating Behavior; Body Image
MeSH Terms: conditions — Feeding Behavior | interventions — Nutrition Assessment; Nutritional Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention schools (educated about nutrition) (Experimental): The research will be conducted in six high schools, three of which are intervention schools . Schools in the district will be divided into 3 layers as 1- Anatolian High Schools, 2- Technical and Vocational High Schools, 3- Imam Hatip High Schools.
  Interventions: Behavioral: Nutrition Education; Behavioral: nutritional status, eating habits
- Control schools (non-educated about nutrition) (Sham Comparator): The research will be conducted in six high schools, three of which are control schools. Schools in the district will be divided into 3 layers as 1- Anatolian High Schools, 2- Technical and Vocational High Schools, 3- Imam Hatip High Schools, and a control school will be determined from each layer by means of a random numbers table
  Interventions: Behavioral: nutritional status, eating habits

INTERVENTIONS:
Behavioral: Nutrition Education — Nutrition interventions consisting of 8 modules (powerpoint supported classroom lesson, video demonstration, role-play, healthy plate model game, poster preparation, bookmarks, refrigerator magnets, etc. preparation of reminder messages, competitions such as slogan-painting contest, activities such as sports and nutrition festival).
  Arms: Intervention schools (educated about nutrition)
Behavioral: nutritional status, eating habits — At the beginning of the study (June 2022), an introductory form (sociodemographic characteristics, body image (Stunkart scale), dietary habits, knowledge about weight status) was applied to all students. Adolescent Nutrition Literacy Scale (ANLS), Instrument of Nutrition Literacy, Mediterranean Diet Quality Index (KID-MED), Eating Attitudes Test 26 (EAT-26), International Physical Activity Questionnaire Short Form (IPAQ) were applied, anthropometric measurements and three-day food consumption records were taken

SUMMARY:
The aim of this study is to determine the effect of nutrition education on nutritional literacy, nutritional status, eating habits and eating behavior in high school students. The research will be conducted in six high schools, three of which are intervention schools and three of which are control schools It is planned that a total of 1000 students will be included in the study from the intervention school and 1000 students from the control school. At the beginning of the study (June 2022), an introductory form (sociodemographic characteristics, body image (Stunkart scale), dietary habits, knowledge about weight status) was applied to all students. Adolescent Nutrition Literacy Scale (ANLS), Instrument of Nutrition Literacy, Mediterranean Diet Quality Index (KID-MED), Eating Attitudes Test 26 (EAT-26), International Physical Activity Questionnaire Short Form (IPAQ) were applied, anthropometric measurements and three-day food consumption records were taken. During the study, nutrition initiatives consisting of 8 modules will be made to the intervention schools. Control schools will not be interfered with during this period.At the end of the study, the procedures applied at the beginning will be repeated.

DETAILED DESCRIPTION:
Lack of knowledge about nutrition is one of the most important causes of nutritional problems. accordingly, wrong eating practices and habits can lead to many complications and health problems. Especially adolescent eating habits form the basis of adult eating habits. The habits acquired during this period can lead to behaviors and attitudes that persist for a long time and are difficult to change.The aim of this study is to determine the effect of nutrition education on nutritional literacy, nutritional status, eating habits and eating behavior in high school students. The research will be conducted in six high schools, three of which are intervention schools and three of which are control schools. Schools in the district will be divided into 3 layers as 1- Anatolian High Schools, 2- Technical and Vocational High Schools, 3- Imam Hatip High Schools, and a control school will be determined from each layer by means of a random numbers table. It is planned that a total of 1000 students will be included in the study from the intervention school and 1000 students from the control school. At the beginning of the study (June 2022), an introductory form (sociodemographic characteristics, body image (Stunkart scale), dietary habits, knowledge about weight status) was applied to all students. Adolescent Nutrition Literacy Scale (ANLS), Instrument of Nutrition Literacy, Mediterranean Diet Quality Index (KID-MED), Eating Attitudes Test 26 (EAT-26), International Physical Activity Questionnaire Short Form (IPAQ) were applied, anthropometric measurements and three-day food consumption records were taken. During the study, nutrition initiatives consisting of 8 modules (powerpoint supported classroom lesson, video demonstration, role-play, healthy plate model game, poster preparation, bookmarks, refrigerator magnets, etc. preparation of reminder messages, competitions such as slogan-painting contest, activities such as sports and nutrition festival) will be made to the intervention schools. Control schools will not be interfered with during this period.At the end of the study, the procedures applied at the beginning (anthropometic measurements, introductory form, scales, food consumption record) will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* studying in the 9th and 10th grades in the selected schools
* agree to participate in the research

Exclusion Criteria:

* Type 1 diabetes
* Metabolic disorders (Phenylketonuria, Maple Syrup Urine Disease, Galactosaemia ect.)
* Pediatric Malabsorption (Celiac, cystic fibrosis, congenital sucrase isomaltase deficiency ect.)
* require a special diet

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1000 (Estimated)
Dates: Start 2022-06-06 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
nutrition literacy | up to 10 months
  To investigate the effects of nutrition education interventions on nutrition literacy. We use Adolescent Nutrition Literacy Scale and Instrument of Nutrition Literacy scale to evaluate the nutrition literacy.
Mediterranean Diet Quality Index (KID-MED) | up to 10 months
  In KIDMED, which is a scale consisting of sixteen questions, each question is answered "Yes" or "No". The scale includes 12 questions about eating habits appropriate for the Mediterranean diet and 4 questions about eating habits not appropriate for the Mediterranean diet. If "Yes" is answered to the questions questioning the eating habits appropriate for the Mediterranean diet, +1 point is obtained, if "Yes" is answered to the questions questioning the eating habits not appropriate for the Mediterranean diet, -1 point is obtained, and 0 point is obtained when no answer is given to the questions. The lowest score that can be obtained from the scale is -4 and the highest score is 12. The total score obtained from the scale is evaluated in three groups as optimal (good) diet quality if it is 8 and above (≥8 points), diet quality that needs to be improved (moderate) if it is between 4-7 points, and very low diet quality (low) if it is 3 and below (≤3 points).
Eating Attitudes Test 26 (EAT-26) | up to 10 months
  It is used to determine whether there is an eating disorder. It is a 6-point Likert-type test consisting of a total of 26 questions. The answers include "always, very often, often, sometimes, rarely, never". A minimum score of "0" and a maximum score of "78" can be obtained from the test. If the test score is above 20, there is a risk of eating behaviour disorder. If the test score is below 20, there is no risk of eating behaviour disorder.
weight and height measurement | up to 10 months
  Height measurement will be made with a portable height meter supported by the wall with light clothes without shoes, with the head upright, looking straight ahead, the line passing through the eyes and ears parallel to the ground, legs straight and closed, arms at the side, shoulders relaxed, heels, hips and shoulders on the Frankfurt plane against the wall.
  Weight measurement will be done with a 100 g sensitive digital scale.
  BMI will be obtained by dividing weight (kg) by the square of height (m), and age and gender appropriate percentile values will be determined. 85-95 percentile will be classified as overweight and ≥95 percentile as obese.
waist circumference measurement | up to 10 months
  Waist circumference will be measured with the help of a non-flexible tape measure, with light clothes, while breathing normally, standing upright, with arms outstretched on both sides, at the point passing through the exact midpoint between the lower ribs and the hip bone.
Food Consumption Record | up to 10 months
  The food consumption record form will be filled in by the researcher for 3 days with 24 hour reminder method. Food and food photo catalogues will be used to determine the measurements and quantities of food consumption. The amount of nutrients included in the meals consumed by the individuals will be calculated using standard recipes. Average energy and nutrient values of the food/drinks consumed will be calculated using the BEBIS programme. In the evaluation of energy and nutrient intakes, recommended daily energy and nutrient values according to gender and age will be used. Accordingly, those who consume ± 50% of the recommended amount of energy and nutrients will be considered adequate (50-150%), and those who consume < 50% will be considered inadequate (50%).
International Physical Activity Questionnaire (IPAQ- Short Form) | up to 10 months
  It was developed by Craig et al. to determine the physical activity status of individuals (Craig et al., 2003). It is a 7-question form whose Turkish validity and reliability was performed by Öztürk (Öztürk, 2005). In this form in which walking, moderate activity, vigorous activity and time spent sitting are questioned, weekly MET values of individuals are calculated and individuals are classified as inactive, minimally active and very active according to the results. A score is obtained as "MET/min/week" by multiplying the minutes, days and MET values of the physical activity performed. In the calculation of the walking score, a walking time of 3.3 METs, 4 METs for moderate physical activity and 8 METs for vigorous physical activity are accepted. If the calculated value is 3000 MET/min/week, it is classified as very active

CONTACTS AND LOCATIONS:
Overall Officials: Murat URHAN, PhD, Principal Investigator — Ege University; Ezgi KARATAŞ, PhD, Principal Investigator — Ege University; Rana N AKDER, Msc, Principal Investigator — Ege University; Ceren AKANALÇI, Msc, Principal Investigator — Ege University; Reci MESERİ, PhD, Principal Investigator — Ege University; Özge KÜÇÜKERDÖNMEZ, PhD, Study Director — Ege University
Locations (1):
- Menemen District Directorate of National Education, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No